CLINICAL TRIAL: NCT05275075
Title: Pilot Trial to Identify microRNAs in Cachexia in Patients With Pancreatic Carcinoma
Brief Title: Identify microRNAs in Cachexia in Pancreatic Carcinoma
Acronym: SCC-miRPanCa
Status: Recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-MIRPANCA
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Resectable Pancreatic Adenocarcinoma
Keywords: pancreatic cancer; cachexia; microRNA; mRNA; PDAC
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — After surgical removal of the pancreatic cancer, part of the tumor tissue will be collected to analyze genes and RNA related to muscle loss in patients with pancreatic tumors. A portion of the tumor will be archived in a repository for future use related to this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic Cancer Cohort: All eligible adenocarcinoma pancreatic cancer patients with operable cancer.
  Interventions: Other: Pancreatic cancer microRNA and messenger RNA expression.

INTERVENTIONS:
Other: Pancreatic cancer microRNA and messenger RNA expression. — Tumor specimens from pancreatic patients will be analyzed for markers associated with muscle loss.

SUMMARY:
The purpose of this study is to determine the proportion of pancreatic patients who experience weight loss and cachexia, and to identify any differences in the genes between patient groups.

DETAILED DESCRIPTION:
This research study will retrospectively examine 1395 patients from the University of Alabama and the University of Oklahoma Stephenson Cancer Center (OU-SCC) pancreatic cancer cohorts. The prospective arm, will enroll a total of 100 eligible volunteers at the OU-SCC. The demographic and medical data from the retrospective and prospective arms will be combined (1495 patients) to ascertain any racial disparities in pancreatic cancer patients with cachexia. Perspective volunteers at the OU-SCC will undergo routine tests to determine if their cancer is operable. Pancreatic tumors will be removed from the eligible patients, as part of their normal standard of care and will be examined for genes that may be related to unexplained muscle loss and compared to tumor tissue from other patients with pancreatic cancer. An optional hand strength exam, and standing on a scale that measures weight, muscle, and body fat will be available to OU-SCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, who is ≥ 18 years old at the time of informed consent.
2. Patients with operable pancreatic tumors diagnosed in the last 12 months prior to consent with clinical discretion or pathology confirmed as adenocarcinoma.
3. Patient has stage I or higher disease who is considered a candidate for surgical resection of pancreatic cancer, with or without neoadjuvant chemotherapy.
4. Ability to provide written informed consent and HIPAA authorization.

Exclusion Criteria:

1. Patients with pancreatic adenocarcinoma who do not meet the criteria for surgical resection.
2. Patient has cancer diagnosis other than primary pancreatic adenocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is inclusive of all races, ethnicities, and gender. Enrollment into the study is restricted to Stephenson Cancer Center site, part of the University Oklahoma Health Sciences Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of African American pancreatic cancer patients with weight loss and cachexia. | 1 - 12 months
  Evaluate weight loss and the markers of cachexia, albumin and psoas cross-sectional area, to see if African Americans with pancreatic cancer patients experience Grade I-IV cachexia at a higher frequency than other racial groups.

SECONDARY OUTCOMES:
Differences in microRNA and messenger RNA tumor expression profiles in all cancer patients undergoing pancreatic surgery. | 1 - 12 months
  Assess fold-change expression differences in microRNA and messenger RNA tumor expression profiles in all cancer patients undergoing pancreatic surgery.
Differences in cachexia-associated RNA signatures in African American pancreatic cancer patients, and other racial groups. | 1 - 12 months
  Assess fold-change expression differences in cachexia-associated RNA signatures in African American pancreatic cancer patients, and other racial groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Jain, MD, Principal Investigator — University of Oklahoma Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No